CLINICAL TRIAL: NCT02591524
Title: Upper and Lower Airway Colonization in Cystic Fibrosis Patients After Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Thomas Fuehner, PD Dr. med. Thomas Fühner, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LuTx-CF-colonization_1
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis; Lungtransplantation; Paranasal Sinus Diseases
MeSH Terms: conditions — Cystic Fibrosis; Paranasal Sinus Diseases | interventions — Nasal Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cystic fibrosis airway colonization (Experimental): Flexible bronchoscopy via the nasal route on the date of baseline visit, nasal lavage at baseline and after 6 month
  Interventions: Other: Bronchoalveolar and Nasal Lavage

INTERVENTIONS:
Other: Bronchoalveolar and Nasal Lavage — A previously scheduled flexible bronchoscopy via the nasal route on the date of baseline visit combined with a nasal lavage and another nasal lavage after 6 month

SUMMARY:
A hot topic in lung transplantation is the treatment of persisting sinus disease/colonization in CF patients to prevent descending graft colonization and chronic allograft dysfunction. From 2012, the Hannover transplantation group has been using a conservative approach with topical nasal inhalation. It is now necessary to analyse the impact of the new approach on graft colonization, incidence of BOS, symptoms, QoL etc in comparison to a historical cohort. It is also important to establish which is the best among the different inhaled antibiotic regimens currently available.

DETAILED DESCRIPTION:
These patients will undergo frequent individual centre based follow up care. At each follow up visit, patients will:

* receive comprehensive clinical examination, history of intercurrent infections and sinus surgery
* receive quantitative assessment, consisting in spirometry (performed according to ATS/ERS guidelines), arterial blood gas analysis, measurement of immunosuppressive drug levels and chest radiographs
* receive questionnaires (quality of life (SNOT-20 GAV), side effects of sinus inhalation, symptom scores)
* be asked to collect a sample of nasal lavage; a sample of BAL (obtained from routinely performed bronchoscopy) will also be collected. These specimens will be analysed for microbiological work up and evaluation of inflammatory markers.

The principle of vibrating inhalation is implemented in novel nebulizers, with which sinonasal inhalation is performed by aerolized medication into one nostril, while the contralateral nostril is occluded and the soft palate elevated as recommended for nasal lavage. The medication is administered into both nostrils for 4-6 min each side during phases of arrest of breathing. Choice of antibiotics depends on resistance testing from microbiological results. Patients will be divided into different groups, on the basis of the inhaled antibiotic regimen being chosen: colistin vs. tobramycin. An alternate therapy with hypertonic saline may be applied to improve sinus clearance. All regimens will be administered with the same machine, i.e. PARI Sinus ™ nebulizer, which, unlike conventional aerosols, allows the deposition of drugs directly into the paranasal sinuses.

The aims of this study are:

* to assess sinus - and pulmonary colonization in cystic fibrosis (CF) lung transplant (LuTx) recipients (frequency of pathogen colonization; load; bacterial species)
* to study association with clinical events (e.g. infections and development of bronchiolitis obliterans syndrome (BOS))
* to develop an optimal inhaled regimen (continuous inhalation/on-off regimen; single or combined antibiotics).
* to compare cohorts receiving sinus surgery in a historical control to a cohort receiving our current conservative strategy (since 2012) of sinonasal vibrating inhalation of antibiotics, in terms of graft colonization, quality of life, overall survival, incidence of chronic lung allograft dysfunction
* to compare inflammatory mediators in upper and lower airway lavages in regard to pathogen colonization, lung function and development of BOS

ELIGIBILITY:
Inclusion Criteria:

* adult (age > 18 yrs)
* cystic fibrosis
* referral for lung transplantation or follow-up after lung transplantation receiving surgical treatment of sinus disease (sinus surgery) or onservative strategy of sinonasal inhalation of antibiotics
* for patients after lung transplantation: needing a previously scheduled flexible bronchoscopy via the nasal route on the date of baseline visit

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
graft colonization after lung Transplantation (lower respiratory tract) | 6 month
  number of patients with positive microbiological testing of bronchoalveolar lavage

SECONDARY OUTCOMES:
Symptoms of rhinosinusitic involvement | 12 month
  symptoms will be assessed with a specific questionnaire (SNOT22_GAV modified)
  * Upper airway colonization with pathogens
  * Incidence of chronic lung allograft dysfunction, infections and hospitalizations
Upper airway colonization with pathogens | 12 month
  number of patients with positive microbiological testing of nasal lavage
Incidence of chronic lung allograft dysfunction, infections and hospitalizations | 12 month
  number of patients with new chronic lung allograft dysfunction, infections and hospitalizations respectivley

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Medizinische Hochschule Hannover, Hanover, Germany